CLINICAL TRIAL: NCT05834192
Title: Comparative Effects of Backward Treadmill Walking and Lower Extremity Cross Training on Gross Motor Function and Balance Among Stroke Patients
Brief Title: Comparative Effects of Backward Treadmill Walking and Lower Extremity Cross Training Among Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0221
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward treadmill walking group (Experimental)
  Interventions: Other: Backward treadmill walking
- Lower extremity cross training (Active Comparator)
  Interventions: Other: Lower extremity cross training

INTERVENTIONS:
Other: Backward treadmill walking — Backward Treadmill walking will be given to this group. Speed settings of treadmill will be established based on the previous motor function of participants. All participants will receive conventional physical exercises which includes general mobility and functional activities. In this study, the 40-minute training programs for both groups will be occur 5 times a week for 6 weeks, with 5 minutes being allocated for warm up, 30 minutes devoted to the main exercise, and 5 minutes for cool down.
  Arms: Backward treadmill walking group
Other: Lower extremity cross training — For cross-training, a strong resistance will be applied by the therapist until a response will be achieved on the contralateral lower extremity at the end range of motion. Resistance will be consistently applied for 10 seconds once a response will be achieved.
  All participants will receive conventional physical exercises which includes general mobility and functional activities. In this study, the 40-minute training programs for both groups will be occur 5 times a week for 6 weeks, with 5 minutes being allocated for warm up, 30 minutes devoted to the main exercise, and 5 minutes for cool down.
  Arms: Lower extremity cross training

SUMMARY:
Stroke is one of the high rated neurological disorders, induced by disruption of brain's blood flow. Stroke can alter the level of consciousness, motor and cognitive skills, sensory perception and language; it all depends on the extent of injury and the region of brain that is affected. Even though all the rehabilitation given to the "stroke" patients, but still 25-30% of the survivors still have gait and balance problem and they require complete physical support before their discharge from the hospital. Backward treadmill walking has reported numerous benefits in improving balance, motor function and gait. Cross training is a technique which is applied to healthy limb of the individual to increase muscle strength and muscle activity.so the aim of this study is to find the effects of backward treadmill walking and lower extremity cross training on gross motor function and balance among stroke patients.

The study will be randomized clinical trials, Participants will be randomly allocated into two groups each group will have 13. This study will be conducted in Safi teaching Hospital Faisalabad. Group A will be treated with backward treadmill walking and group B will be treated with lower extremity cross training. All participants will receive conventional physical exercises which includes general mobility and functional activities. In this study, the 40-minute training programs for both groups will be occur 5 times a week for 6 weeks, with 5 minutes being allocated for warm up, 30 minutes devoted to the main exercise, and 5 minutes for cool down. Outcome will be measured before and after giving treatment by using Tinetti performance oriented mobility assessment and lower extremity functional scale. The results will be calculated by using SPSS version 25. Frequencies and mean standard deviation will be measured, parametric and non-parametric tests will be applied

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patient diagnosed within last 6 months to 1 year
* Age 55 to 75 years
* Cognition score on Mini-mental state examination > 24
* Able to independently walk 10 m without walking aids
* Able to understand instructions

Exclusion Criteria:

* Who will have visual or vestibular injury
* Patients having history of orthopedic surgery or having an orthopedic condition
* Who will have >grade 2 on modified Ashworth Scale (MAS)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | 8 weeks
  It consists of 20 questions designed to assess a person's ability to perform everyday tasks, such as getting into or out of the bath, walking between rooms, squatting, and sitting for 1 hour. Performance is rated on a 5-point scale with maximum score of 80. Lower score shows greater disability
Tinetti Performance Oriented Mobility Assessment (POMA) | 8 weeks
  it comprises 16 items (9 balance-related and 7 gait-related items). The highest achievable score being 28 points (16 for balance and 12 for gait). A higher score indicates better balance. A cutoff score greater than 17 points has been associated with fall risk in the older adult population.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, Masters, Principal Investigator — Riphah International University
Locations (1):
- Safi teaching hospital Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No